CLINICAL TRIAL: NCT06782334
Title: Phase 1/2 Study of AMT-116 in Patients with Advanced Solid Tumors
Brief Title: AMT-116 in Patients with Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Multitude Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AMT-116-02
Record Dates: First submitted 2024-12-20; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Phase I: Dose escalation (Experimental): Five dose levels in the Phase I part of the study
  Interventions: Drug: AMT-116
- Phase II: Dose Expansion (Other): Patients in phase II will be enrolled based on the RP2D (Recommended Phase 2 Dose) determined from phase I dose escalation data.
  Interventions: Drug: AMT-116

INTERVENTIONS:
Drug: AMT-116 — AMT-116 is an antibody Drug Conjugate (ADC)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of AMT-116 monotherapy in subjects with advanced solid tumors. The study is divided into two parts: the part I is dose escalation and the Part Ⅱ for expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be willing and able to sign the ICF, and to adhere to the study visit schedule and other protocol requirements.
2. Age ≥18 years (at the time consent is obtained).
3. Patients with histologically confirmed, unresectable advanced solid tumor. Preferred tumor types include non-small cell lung, head and neck, esophageal, cervical, breast, bladder, gastric, biliary tract, skin squamous cell, liver, and basal cell cancer.
4. Patients who have undergone at least one systemic therapy and have radiologically or clinically determined progressive disease during or after most recent line of therapy, and for whom no further standard therapy is available, or who are intolerable to standard therapy.
5. Patients must have at least one measurable lesion as per RECIST version 1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
7. The anticipated survival duration is no less than three months.
8. Patients must have adequate organ function
9. Women of child-bearing potential (WCBP) must consent to the use of two effective contraceptive methods during the study treatment period and for at least 12 weeks after the final administration of IMP
10. Women of child-bearing potential (WCBP) must have a negative serum pregnancy test within seven days preceding the initial administration of the investigational medicinal product (IMP).
11. Male patients must agree to use a latex condom, even if they had a successful vasectomy, while on study treatment and for at least 12 weeks after the last dose of the IMP.
12. Male patients must agree not to donate sperm, and female patients must agree not to donate eggs, while on study treatment and for at least 12 weeks after the last dose of the IMP.
13. Availability of tumour tissue sample (either an archival specimen or a fresh biopsy material) at screening.

Exclusion Criteria:

1. Prior therapy with ADC based on Top1 inhibitor.
2. Central nervous system (CNS) metastasis.
3. Active or chronic skin disorder requiring systemic therapy.
4. History of Steven's Johnson's syndrome or Toxic Epidermal Necrolysis syndrome.
5. Active ocular conditions requiring treatment or close monitoring, including, but not limited to: macular degeneration, papilledema, active diabetic retinopathy with macular oedema, wet age-related macular degeneration requiring intravitreal injections, or uncontrolled glaucoma.
6. Persistent toxicities from previous systemic anti-neoplastic treatments of Grade >1.
7. Systemic anti-neoplastic therapy within five half-lives or 21 days, whichever is shorter, prior to first dose of the IMP.
8. Radiotherapy to lung field at a total radiation dose of ≥20 Gy within 6 months, wide-field radiotherapy (e.g., > 30% of marrow-bearing bones) within 28 days.
9. Major surgery (not including placement of vascular access device or tumor biopsies) within 28 days prior to the first dose of the IMP, or no recovery from side effects of such intervention.
10. Significant cardiac disease, such as recent (within six months prior to first dose of the IMP) myocardial infarction or acute coronary syndromes (including unstable angina pectoris), congestive heart failure (New York Heart Association class III or IV), uncontrolled hypertension, uncontrolled cardiac arrhythmias.
11. Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, or current ILD/pneumonitis, or suspected ILD/pneumonitis (e.g., idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, etc.).
12. History of thromboembolic or cerebrovascular events, including transient ischemic attacks, cerebrovascular accidents, deep vein thrombosis, or pulmonary emboli within six months prior to first dose of the IMP.
13. Acute and/or clinically significant bacterial, fungal or viral infection including hepatitis B virus (HBV), hepatitis C virus (HCV), and known human immunodeficiency virus (HIV).
14. Administration of a live vaccine within 28 days prior to the administration of the first dose of the IMP.
15. Patients requiring concurrent treatment of strong inhibitors or inducers of cytochrome P450 3A4 enzyme (CYP3A4) within 2 weeks prior to the first dose and during the study treatment.
16. Known or suspected severe allergy/hypersensitivity (resulting in treatment discontinuation) to monoclonal antibodies.
17. Known or suspected intolerance to the components of the IMP.
18. Concurrent participation in another investigational therapeutic clinical trial.
19. Patients with known active alcohol or drug abuse.
20. Pregnant or breast-feeding females.
21. Mental or medical disorders that prevent patients from signing informed consent or complying with the study, or other severe acute or chronic medical or psychiatric disorders or abnormal laboratory results that may increase the risk associated with study participation or IMP administration or may interfere with the interpretation of study results and, in the investigator's judgment, make patients ineligible for enrollment in the study.
22. There was a history of malignant tumors other than the selected diagnosis within 5 years prior to the first administration of IMP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Phase I: Maximum Tolerated Dose(MTD) and the Recommended Phase 2 Dose(RP2D) of AMT-116 | approximately 12 months
  The MTD（Maximum Tolerated Dose） and RP2D（Recommended Phase 2 Dose） will be determined for expansion using dose limiting toxicities (DLTs) and all other available study data
Phase I: Type, incidence and severity of Adverse Events,Dose Limiting Toxicities (DLTs) | approximately 12 months
  Assess safety and tolerability of AMT-116 by the National Cancer Institute (NCI) Common Terminology Criteria for AEs (CTCAE) version 5.0
Phase II: Objective Response Rate(ORR) | approximately 18 months
  To evaluate the objective response rate (ORR) [Complete Response (CR) + Partial Response (PR)] according to the RECIST v1.1
Phase II: Type, incidence and severity of Adverse Events | approximately 18 months
  Assess safety and tolerability of AMT-116 by the National Cancer Institute (NCI) Common Terminology Criteria for AEs (CTCAE) version 5.0

SECONDARY OUTCOMES:
Phase I: Overall Response Rate (ORR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | approximately 12 months
  Proportion of patients achieving Complete Response (CR) or Partial Response (PR)
Phase I Disease Control Rate (DCR) according to the RECIST v1.1 | approximately 12 months
  Proportion of patients achieving CR, PR or Stable Disease (SD)
Phase I: Progression-free Survival (PFS) | approximately 12 months
  Time from date of start of treatment to date of the first progression or death, whichever occurs first
Phase I: Levels of target expression or Tumor Infiltrating Lymphocyte in tumor tissue | approximately 12 months
  To assess levels of target expression and Tumor Infiltrating Lymphocyte in tumor tissue
Phase I: Concentration of anti-drug antibodies (ADA) | approximately 12 months
  Immunogenicity profile characterized by concentration of ADAs
Phase I: Maximum observed concentration (C[max]) | approximately 12 months
  Pharmacokinetic profile characterized by the maximum observed concentration (C[max]) of AMT-116
Phase I: Area under the curve (AUC) | approximately 12 months
  Pharmacokinetic profile characterized by the area under the curve (AUC) of AMT-116
Phase I: Terminal half-life (t[1/2]) | approximately 12 months
  Pharmacokinetic profile characterized by the terminal half-life (t[1/2]) of AMT-116
Phase I: Time to maximum concentration (Tmax) | approximately 12 months
  Pharmacokinetic profile characterized by the time to maximum concentration (Tmax) of AMT-116
Phase II: Disease Control Rate (DCR) according to the RECIST v1.1 | approximately 18 months
  Proportion of patients achieving CR, PR or Stable Disease (SD)
Phase II: Progression-free Survival (PFS) according to RECIST v1.1 | approximately 18 months
  Time from date of start of treatment to date of the first progression or death, whichever occurs first.
Phase II: Duration of response (DOR) | approximately 18 months
  DOR is defined as the time from the date of first documented CR or PR to PD or death due to any cause, whichever occurs first.
Phase II: Time to response(TTR) | approximately 18 months
  The time from the start date of treatment to the date of the first response assessment (PR or CR)
Phase II: Levels of target expression in tumor tissue | approximately 18 months
  To assess levels of target expression in tumor tissue and correlation of those levels with responses and toxicity.
Phase II: Percentage of patients with ADA formation to AMT-116. | approximately 18 months
  To obtain Percentage of patients with ADA formation to AMT-116
Phase II: Maximum observed concentration (C[max]) | approximately 18 months
  To characterize the PK profile of AMT-116 by analyzing maximum observed concentration (C[max]) of the ADC, total antibody, and free payload.
Phase II: Area under the curve (AUC) | approximately 18 months
  To characterize the PK profile of AMT-116 by analyzing area under the curve (AUC) of the ADC, total antibody, and free payload.
Phase II: Terminal half-life (t[1/2]) | approximately 18 months
  To characterize the PK profile of AMT-116 by analyzing the pharmacokinetic parameter Terminal half-life (t½ )of the ADC, total antibody, and free payload.
Phase II: Time to maximum concentration (Tmax) | approximately 18 months
  To characterize the PK profile of AMT-116 by analyzing the pharmacokinetic parameter time to maximum concentration (Tmax) of the ADC, total antibody, and free payload.

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Zhujiang Hospital of Southern Medical University(The Second Clinical Medical College), Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Hunan Cancer Hospital, Changsha, Hunan
  - Zhejiang cancer hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital and Yuying Childrens Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No